CLINICAL TRIAL: NCT03091777
Title: A Multicenter, Randomized, Double-Blind, Vehicle Controlled Study Evaluating the Therapeutic Equivalence and Safety of GDC-229 (Investigational Metronidazole 0.75% Vaginal Gel) and Metronidazole 0.75% Vaginal Gel in the Treatment of Bacterial Vaginosis
Brief Title: Study Evaluating the Equivalence of GDC-229 and Metronidazole Vaginal Gel 0.75% in the Treatment of Bacterial Vaginosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Balmoral Medical company (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDC-229-002
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Results first posted 2019-10-14 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-09

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; vaginal infection; BV
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Drug (Experimental): GDC-229 gel applied vaginally as directed.
  Interventions: Drug: GDC-229
- Reference Drug (Active Comparator): Metronidazole Vaginal Gel, 0.75% applied vaginally as directed.
  Interventions: Drug: Metronidazole Vaginal Gel 0.75%
- Vehicle Placebo Gel (Placebo Comparator): GDC-229 Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GDC-229 — GDC-229 is a vaginal gel.
  Arms: Test Drug
Drug: Metronidazole Vaginal Gel 0.75% — Metronidazole Vaginal Gel 0.75% is an FDA-approved drug
  Arms: Reference Drug
Drug: Placebo — Inactive arm of the study
  Arms: Vehicle Placebo Gel

SUMMARY:
This research study is being done to compare the safety and efficacy of GDC-229 (test drug) against the currently marketed reference drug (metronidazole 0.75% vaginal gel) and to establish that these two drugs work better than placebo in subjects with BV.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant female aged ≥ 18 years who is in good general health
2. Diagnosis of BV
3. Willing to refrain from using any intravaginal product (e.g., spermicide, tampon, douche, feminine deodorant spray, diaphragm, vaginal ring birth control, or condom with spermicide or insertion into the vagina of any drug or non-drug product during treatment), other than study treatment for the duration of the trial
4. Subjects of childbearing potential who have a negative urine pregnancy test at the Entry Visit (Visit 1) and agree to use an acceptable form of birth control throughout the study
5. Able to understand and willing to sign the informed consent form (ICF) and able to comply with the requirements of the protocol

Exclusion Criteria:

1. History of alcohol or substance abuse
2. Experienced a clinically significant medical event within 90 days
3. Abnormal pap or high risk human papillomavirus (HPV)
4. History or presence of clinically significant central nervous system (CNS), cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, gynecologic, dermatologic, neurologic, oncologic, or psychiatric disease
5. Pregnant, lactating, or planning to become pregnant or breastfeed during the study period
6. Primary or secondary immunodeficiency
7. Evidence of any vulvovaginitis at screening other than BV
8. History of hypersensitivity or allergy to metronidazole, parabens, other nitroimidazole derivatives, or other ingredients of the GDC 229 (metronidazole 0.75% vaginal gel), metronidazole 0.75% vaginal gel (Oceanside Pharmaceuticals), or vehicle gel
9. Participating in another clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Non-pregnant female aged ≥ 18 years who is in good general health
Enrollment: 871 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 103, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2017 to November 2017
  The location of clinical sites included women's health clinics and clinical research centers
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Period: Overall Study
Arm/Group | Test Drug | Reference Drug | Vehicle Placebo Gel
Started | 289 | 288 | 294
Completed | 257 | 255 | 257
Not Completed | 32 | 33 | 37
Not completed — Pregnancy | 2 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 4
Not completed — Withdrawal by Subject | 4 | 2 | 6
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Lost to Follow-up | 12 | 14 | 7
Not completed — Lack of Efficacy | 0 | 0 | 5
Not completed — Noncompliance with study drug | 2 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Abnormal Laboratory Value | 7 | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Drug | Reference Drug | Vehicle Placebo Gel | Total
Number analyzed (Participants) | 287 | 285 | 292 | 864
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (8.56) | 33.2 (9.61) | 33.5 (9.77) | 33.3 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 285 | 292 | 864
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 50 | 56 | 160
  Not Hispanic or Latino | 233 | 233 | 235 | 701
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 4
  Asian | 1 | 4 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 161 | 158 | 164 | 483
  White | 117 | 117 | 117 | 351
  More than one race | 2 | 1 | 3 | 6
  Unknown or Not Reported | 4 | 4 | 2 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 287 | 285 | 292 | 864

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure
Description: Resolution of clinical signs and symptoms
Time Frame: Day 21-30
Population: Modified Intent-to-Treat (mITT) population: All randomized subjects who received study treatment and returned for at least one post-baseline visit, but excluding those who demonstrate a positive test result for other concomitant vaginal or cervical infections at baseline (e.g. C. trachomatis, N. gonorrhoeae) or who have a baseline Nugent score<4.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Drug | Reference Drug | Vehicle Placebo Gel
Number analyzed (Participants) | 245 | 245 | 243
Participants | 135 | 129 | 74
Statistical Analysis 1: Comparison: Test Drug vs Vehicle Placebo Gel; Test type: Superiority; p < 0.001, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Reference Drug vs Vehicle Placebo Gel; Test type: Superiority; p < 0.001, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 21 months
Arm/Group | Test Drug | Reference Drug | Vehicle Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/287 | 0/285 | 0/292
Serious Adverse Events (participants affected / at risk) | 2/287 | 0/285 | 2/292
Other Adverse Events (participants affected / at risk) | 44/287 | 37/285 | 35/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Drug (N=287) | Reference Drug (N=285) | Vehicle Placebo Gel (N=292)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Enterocolic Intussusception
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — Acute Cholecystitis
Sickle Cell Anaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) — Worsening Sickle Cell Anemia
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Exacerbation Of Supraventricular Tachycardia
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Drug (N=287) | Reference Drug (N=285) | Vehicle Placebo Gel (N=292)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (3)
Trichomoniasis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Vulvovaginal candidiasis (Infections and infestations) | 15 (15) | 10 (10) | 12 (12)
Vulvovaginal mycotic infection (Infections and infestations) | 13 (13) | 17 (17) | 10 (10)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03091777/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT03091777/SAP_001.pdf